CLINICAL TRIAL: NCT01517971
Title: Validation of Molecular Prognostic Tests in NSCLC
Brief Title: Studying Tumor Tissue Samples From Patients With Early-Stage Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150807; CALGB-150807; CDR0000720368 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative (whole-genome expression): RNA extracted from archived tumor tissue samples are analyzed for whole-genome expression profiling by Gene Profiling Array cGMP U133 P2 and RT-PCR.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in predicting the risk of cancer returning after surgery in tissue samples of patients with early-stage non-small cell lung cancer. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer and predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and validate a clinically useful molecular prognostic signature based on ribonucleic acid (RNA)-expression arrays to accurately distinguish between good and poor outcome in patients with stage 1B non-small cell lung cancer (NSCLC) (T2aN0M0) by predicting the risk of cancer recurrence after surgery.

SECONDARY OBJECTIVES:

I. To develop and validate a clinically useful prognostic signature for stage 1A NSCLC (T1a-bN0M0) that accurately predicts the risk of post-operative cancer recurrence and is part of a prognostic classifier, which also includes histological, pathological, and demographic parameters as in the primary objective.

II. To determine the effects on test accuracy of the histological subtype (adenocarcinoma [AC] vs squamous cell [SQA]) for each of the stage specific prognostic classifiers.

III. To determine the relevant statistical features, including accuracy of predicting overall survival, cancer specific survival, and disease free survival at 3 and 5 years, for each of the prognostic classifiers validated.

IV. To utilize the validated prognostic signatures and classifiers in stage 1B NSCLC to determine whether these can reliably predict good outcome among stage II NSCLC patients.

OUTLINE:

RNA extracted from archived tumor tissue samples are analyzed for whole-genome expression by Affymetrix microarrays (Gene Profiling Array cGMP U133 P2) and reverse transcriptase-polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Registration to CALGB-140202
* The subject population to be studied in this protocol includes patients selected from CALGB-140202; all such patients have signed a written informed consent document meeting all federal, state and institutional guidelines as part of entry into that trial; the CALGB does not require that a separate consent form be signed for this study
* All samples to be studied were obtained and stored as part of CALGB-140202; the material and data obtained from the patient's protocol record will be used to obtain appropriate clinical information; in no instance will the patient be contacted directly
* Tumor specimens need to have 40% tumor content to be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NSCLC enrolled on the Cancer and Leukemia Group B (CALGB) 140202
Sampling Method: Probability Sample
Enrollment: 1060 (Actual)
Dates: Start 2012-01; Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Recurrence | up to 36 months

SECONDARY OUTCOMES:
Cancer specific survival | Up to 36 months
Disease-free survival | up to 36 months
Overall survival | up to 36 months
Probability of death due to other causes | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, MD, Study Chair — Brigham and Women's Cancer Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bueno R, Richards WG, Harpole DH, Ballman KV, Tsao MS, Chen Z, Wang X, Chen G, Chirieac LR, Chui MH, Franklin WA, Giordano TJ, Govindan R, Joshi MB, Merrick DT, Rivard CJ, Sporn T, van Bokhoven A, Yu H, Shepherd FA, Watson MA, Beer DG, Hirsch FR. Multi-Institutional Prospective Validation of Prognostic mRNA Signatures in Early Stage Squamous Lung Cancer (Alliance). J Thorac Oncol. 2020 Nov;15(11):1748-1757. doi: 10.1016/j.jtho.2020.07.005. Epub 2020 Jul 24. PMID 32717408